CLINICAL TRIAL: NCT06044233
Title: A Randomized, Open, Two-sequence, Two-cycle, Double-cross Design Bioequivalence Trial of Fasting Single Oral STI-1558 Capsule in Healthy Chinese Subjects
Brief Title: A Bioequivalence Trial of Fasting Single Oral STI-1558 Capsule in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zhejiang ACEA Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MPR-COV-105CN
Record Dates: First submitted 2023-09-15; First posted 2023-09-21 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — STI-1558

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR group (Experimental): Subjects in the TR group will take the test preparation (T) 200 mg/ pill × 1 pill on day 1 (D1) and the reference preparation (R) 200 mg/ pill × 1 pill on day 8 (D8).
  Interventions: Drug: STI-1558
- RT group (Experimental): Subjects in the RT group will take the reference preparation (R) 200 mg/ pill × 1 pill on day 1 (D1) and the test preparation (T) 200 mg/ pill × 1 pill on day 8 (D8).
  Interventions: Drug: STI-1558

INTERVENTIONS:
Drug: STI-1558 — STI-1558 test preparation and reference preparation
  Other Names: An oral small molecule prodrug that effectively inhibits the SARS-CoV-2 main protease (Mpro).

SUMMARY:
This study is a randomized, open, single-dose, two-sequence, two-cycle, double-cross design bioequivalence study.

32 eligible subjects will be randomly assigned to TR group and RT group in a 1:1 ratio. Subjects in the TR group will take the test preparation (T) 200 mg/ pill × 1 pill on day 1 (D1) and the reference preparation (R) 200 mg/ pill × 1 pill on day 8 (D8). The sequence of medication in RT group is reversed from TR group. Wash for at least 7 days between doses.

Screening was performed within 28 days prior to initial dosing, and all eligible subjects were admitted to the clinical research Center 1 day prior to Cycle 1 dosing (D-1) and discharged on day 10 of the study (D10) after completing Cycle 2 PK blood collection, corresponding safety examination, and evaluation. On the 14th day of the study (± 1 day), the clinical research center was returned for follow-up to further evaluate the safety and tolerability of the subjects.

DETAILED DESCRIPTION:
This study is a randomized, open, single-dose, two-sequence, two-cycle, double-cross design bioequivalence study.

32 eligible subjects will be randomly assigned to TR group and RT group in a 1:1 ratio. Subjects in the TR group will take the test preparation (T) 200 mg/ pill × 1 pill on day 1 (D1) and the reference preparation (R) 200 mg/ pill × 1 pill on day 8 (D8). The sequence of medication in RT group is reversed from TR group. Wash for at least 7 days between doses.

The trial drug STI-1558 should be taken with approximately 240 ml of water after fasting overnight for at least 10h. Except for drinking water, water should be prohibited for at least 1h before and after administration, and fasting should be at least 4h after administration. Test drugs (T and R) must be swallowed whole and not chewed, crushed or separated. In order to ensure the subject's compliance with the medication procedure, the staff should check the subject's mouth after taking the medication.

Screening was performed within 28 days prior to initial dosing, and all eligible subjects were admitted to the clinical research Center 1 day prior to Cycle 1 dosing (D-1) and discharged on day 10 of the study (D10) after completing Cycle 2 PK blood collection, corresponding safety examination, and evaluation. On the 14th day of the study (± 1 day), the clinical research center was returned for follow-up to further evaluate the safety and tolerability of the subjects.

ELIGIBILITY:
Inclusion Criteria:

1. The subject fully understands the purpose, nature, method and possible adverse reactions of the test, voluntarily becomes a participant, and signs an informed consent form (ICF) before the start of any procedure;
2. Healthy adult males or females aged 18-45 years (including the threshold) at the time of signing the ICF;
3. At the time of signing the ICF and on the day of hospitalization, the body mass index (BMI) is 19-24 kg/m2 (including the threshold), and the weight is not less than 45 kg for women and not less than 50 kg for men;
4. Good health with normal or abnormal results of history, vital signs, physical examination, 12-lead ECG, laboratory tests (blood routine, blood glucose, blood biochemistry, urine routine and coagulation tests) and hemodialysis during the screening period (NCS);
5. Fertile Women (WOCBP) subjects must consent to the use of one or more effective contraceptive methods from the screening period to 30 days after the last dose;
6. Fertile male subjects must consent to the use of one or more effective contraceptive methods within 30 days from the first dose to the last dose;
7. The subject is able to communicate well with the investigator (or designee) and understands and complies with the requirements of the study.

Exclusion Criteria:

1. Patients who have difficulty in venous blood collection or have a history of needle fainting or blood fainting;
2. Pregnant or lactating;
3. Allergic constitution or allergic to any ingredient in STI-1558 capsule preparation;
4. Within 1 month prior to screening or within 5 half-lives of the drug (subject to older age) and those who have been enrolled in other clinical trials (including but not limited to investigational drugs, vaccines, biologics, devices, blood products, etc.);
5. Have a history of gastrointestinal (such as duodenal ulcer, gastrointestinal bleeding), liver or kidney related, or other medical history that the investigator (or his designee) determines may affect the absorption, distribution, metabolism, and excretion of oral drugs;
6. Have any clinical history of serious diseases (including but not limited to respiratory system, circulatory system, digestive system, blood system, endocrine system, immune system, skin and mucosal system, psychiatric nervous system, ent department and other related diseases);
7. Those who underwent major surgery within 3 months prior to screening, or did not fully recover from surgery, or planned to have surgery during the study period;
8. Within 14 days prior to screening and screening of patients with a history of fever;
9. QT interval prolongation: QTcF > 450 msec (male); QTcF > 470 msec (female);
10. Those who were vaccinated within 14 days prior to screening and those who were screened until check-in or planned to be vaccinated during the study period;
11. Within 7 days before screening and screening of patients who have used BCRP substrate drugs;
12. Those who have used CYP3A4 inhibitor, strong inducer, or CYP1A2 inhibitor within 7 days prior to screening and those who have been screened;
13. Within 14 days prior to screening or within 5 half-lives of the drug (whichever is older), and to those who have been admitted to use any other prescription, over-the-counter or Chinese herbal medicine (other than contraceptive drugs or topical drugs assessed by the investigator to be applicable);
14. Had a history of drug abuse within 2 years prior to screening, or tested positive for drug abuse upon admission (D-1);
15. Patients with a history of blood donation or blood loss (excluding female menstrual blood loss) exceeding 400 mL within 3 months before screening;
16. Those who consumed more than 14 units of alcohol per week in the 3 months prior to screening (1 unit of alcohol =360 mL beer or 45 mL spirits with 40% alcohol or 150 mL wine), or had consumed alcoholic products within 48 hours prior to the first dose, or were unable to abstinent during the study period, or tested positive for alcohol breath test at admission (D-1);
17. Smokers who smoked more than 5 cigarettes per day in the 3 months before screening, or who could not guarantee no smoking during the trial period;
18. Excessive consumption of tea, coffee or caffeinated beverages (defined as: at least 8 cups per day, 1 cup =250 ml) in the 3 months prior to screening, or intake of caffeine or xanthine-rich foods or beverages (such as coffee, tea, chocolate, cola, etc.) within 48 hours prior to the first dose;
19. Consumed food, juice or drink containing grapefruit, lime, cinchona peel or quinine within 48 hours before screening and until check-in;
20. Positive or above the upper limit of the reference range for four hemodialysis tests, including hepatitis B surface antigen (HBsAg), hepatitis C (HCV) antibodies, human immunodeficiency virus (HIV) antibodies or treponema pallidum antibodies;
21. Other circumstances in which the investigator (or his designee) deems it inappropriate to participate in the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Comparison of maximum observed concentration(Cmax) profiles of two different kinds of oral STI-1558 to determine the Relative Bioavailability | Up to 2 weeks
  To compare Cmax of the test preparation (T) 200 mg/ pill × 1 pill on day 1 (D1) and the reference preparation (R) 200 mg/ pill × 1 pill on day 8 (D8) in healthy adult , human subjects under fasting conditions, to establish relative bioavailability.
Comparison of Area Under the Curve (AUC) from time 0 to last time point(AUC0-t) profiles of two different kinds of oral STI-1558 to determine the Relative Bioavailability | Up to 2 weeks
  To compare AUC0-t of the test preparation (T) 200 mg/ pill × 1 pill on day 1 (D1) and the reference preparation (R) 200 mg/ pill × 1 pill on day 8 (D8) in healthy adult , human subjects under fasting conditions, to establish relative bioavailability.
Comparison of AUC from time 0 extrapolated to infinity(AUC0-inf ) profiles of two different kinds of oral STI-1558 to determine the Relative Bioavailability | Up to 2 weeks
  To compare AUC0-inf of the test preparation (T) 200 mg/ pill × 1 pill on day 1 (D1) and the reference preparation (R) 200 mg/ pill × 1 pill on day 8 (D8) in healthy adult , human subjects under fasting conditions, to establish relative bioavailability.

SECONDARY OUTCOMES:
Comparison of Tmax of two different kinds of oral STI-1558 to determine the Relative Bioavailability | Up to 2 weeks
  To compare Tmax of the test preparation (T) 200 mg/ pill × 1 pill on day 1 (D1) and the reference preparation (R) 200 mg/ pill × 1 pill on day 8 (D8) in healthy adult , human subjects under fasting conditions, to establish relative bioavailability.
Comparison of t1/2 of two different kinds of oral STI-1558 to determine the Relative Bioavailability | Up to 2 weeks
  To compare t1/2 of the test preparation (T) 200 mg/ pill × 1 pill on day 1 (D1) and the reference preparation (R) 200 mg/ pill × 1 pill on day 8 (D8) in healthy adult , human subjects under fasting conditions, to establish relative bioavailability.
Comparison of λz of two different kinds of oral STI-1558 to determine the Relative Bioavailability | Up to 2 weeks
  To compare λz of the test preparation (T) 200 mg/ pill × 1 pill on day 1 (D1) and the reference preparation (R) 200 mg/ pill × 1 pill on day 8 (D8) in healthy adult , human subjects under fasting conditions, to establish relative bioavailability.
Comparison of %AUCex of two different kinds of oral STI-1558 to determine the Relative Bioavailability | Up to 2 weeks
  To compare %AUCex of the test preparation (T) 200 mg/ pill × 1 pill on day 1 (D1) and the reference preparation (R) 200 mg/ pill × 1 pill on day 8 (D8) in healthy adult , human subjects under fasting conditions, to establish relative bioavailability.

CONTACTS AND LOCATIONS:
Overall Officials: Chen Jian, master, Study Chair — Zhejiang Hospital
Locations (1):
- Zhejiang Xiaoshan Hospital, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No